CLINICAL TRIAL: NCT01478399
Title: Phase 1 Open-Label Pharmacokinetic, Safety and Tolerability Study of a Single Subcutaneous Dose of Glymera (PB1023) Injection in Subjects With Normal Renal Function and Subjects With Impaired Renal Function
Brief Title: Pharmacokinetic, Safety/Tolerability Study of a Single SC Dose of PB1023 Injection in Subjects With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB1023-PT-CL-0003
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Impaired Renal Function (Experimental): Subjects have impaired renal function matched to subjects with normal renal function by age and weight.
  Interventions: Drug: PB1023 Injection
- Normal Renal Function (Experimental): Subjects have normal renal function matched to subjects with impaired renal function by age and weight.
  Interventions: Drug: PB1023 Injection

INTERVENTIONS:
Drug: PB1023 Injection — 90 mg Dose

SUMMARY:
Primary objective:

To compare the pharmacokinetic profile of Glymera (PB1023) Injection after a single dose administered by subcutaneous injection to subjects with normal renal function and impaired renal function.

Secondary objectives:

To evaluate the safety and tolerability of Glymera (PB1023) Injection administered as a subcutaneous injection in adult subjects with normal renal function and impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 - 79 years of age inclusive.
* BMI 19 - 40 kg/m2.
* Renally Impaired Subjects: In otherwise stable health except for Renal Disease.
* Healthy volunteers must have/be: eGFR as calculated by MDRD of ≥ 80 mL/min, and Matched to renally impaired subjects for age (± 15 years), weight (± 15 kg), and if possible BMI, race and gender.
* Subjects with renal impairment must have 2 separate eGFR that are within 20% of each other and clinically stable for a minimum of 6 months.
* No clinically relevant abnormalities in the results of the laboratory screening or admission evaluation other than those consistent with renal impairment or related disease/disorder in the appropriate subject group as determined by the Investigator.

Exclusion Criteria:

* Currently taking or have taken a GLP -1 agent (e.g., Byetta®, Victoza®) within the past year.
* Subjects who have previously received PB1023.
* Known allergy or serious adverse effect to an approved or investigational GLP-1 receptor analog/agonist.
* Serious Infection within 60 days of admission.
* Donation or loss of greater than 400 mL of blood 56 days prior to enrollment.
* Unstable cardiovascular disease defined as per protocol.
* Clinically significant hepatic dysfunction defined as per protocol.
* Female subjects who are pregnant, trying to become pregnant or lactating.
* Known history of or active alcohol or drug abuse within 12 months prior to Screening or positive alcohol and/or drug screen.
* Positive for Human Immunodeficiency Virus (HIV) antibodies, Hepatitis B surface antigen (HBsAg) or Hepatitis C Virus (HCV) antibodies.
* Participating in any other study at time of screening other than observational studies or have received any other investigational drug or device within 30 days or 5 half-lives prior to dosing or are taking part in a non-drug study which in the opinion of the Investigator would interfere with the outcome of the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Pre-Dose, 1, 4, 8 and 12 hours post-dose, Day 1, 2, 3, 5, 7, 10, 14, 21 and 28
  The PK analysis population will consist of subjects that complete the study and have sufficient data for PK analysis. The following parameters will be evaluated: t1/2, AUC(0-inf), Tmax, Cmax, elimination rate constant, CL/F, Vz/F.

SECONDARY OUTCOMES:
Safety/Tolerability | Screening to Final Visit (Approximately 6 weeks)
  Safety and tolerability will be evaluated by analyses of the incidence of adverse events. Vital signs, ECGs and safety laboratory parameters will be presented descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K. Ries, MD, Principal Investigator — Prism Research Inc.
Locations (2):
- United States (2):
  - Prism Research, Saint Paul, Minnesota
  - New Orleans Center for Clinical Research, Knoxville, Tennessee